CLINICAL TRIAL: NCT03088449
Title: Investigation of the Clinical,Serological and Genetic Factors That Determine Primary Non-response, Loss of Response and Adverse Drug Reactions to Anti-TNF Drugs in Patients With Active Luminal Crohn's Disease
Brief Title: Personalising Anti-TNF Therapy in Crohns Disease (PANTS)
Acronym: PANTS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Royal Devon and Exeter NHS Foundation Trust (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); AbbVie (Industry); Pfizer (Industry); Centre for Ocular Research & Education, Canada (Other); Napp Pharmaceuticals Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: RDE 1307805
Record Dates: First submitted 2014-01-06; First posted 2017-03-23 (Actual); Last update posted 2018-06-21 (Actual); Status verified 2018-06

CONDITIONS: Crohn Disease
Keywords: Crohns disease; primary non response; lose of response; personalising anti-TNF therapy; Anti-TNF; PANTS; Biosimilars
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA, RNA, STOOL, SERUM will be collected over the 3 years period from multiple time points.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To develop a cost-effective, individualised anti-TNF treatment strategy for patients with Crohn's disease which maximizes benefit and minimises harm.

The primary objective of this study is to investigate the mechanisms that underlie primary non-response (PNR), loss of response (LOR) and adverse drug reactions (ADRs) to anti-TNF drugs in patients with active luminal Crohn's disease.

DETAILED DESCRIPTION:
This is a prospective uncontrolled cohort study investigating primary non-response (PNR), loss of response (LOR) and adverse drug reactions (ADR) to IFX and ADA in patients with severe active luminal Crohn's disease. The primary objective of this study is to investigate the mechanisms that underlie PNR, LOR, ADRs and remission after anti-TNF withdrawal. The secondary aims are to develop personalised anti-TNF treatment strategies, through the identification of clinically meaningful serological and genetic predictive markers.

This study builds on the achievements of the UK and international IBDGC in identifying IBD susceptibility genes. These discoveries have provided important insights into disease pathogenesis but are not expected to have an impact in the clinic for a number of years. This study aims to take genetics and biomarker discovery into the IBD clinic to address questions of immediate clinical importance.

The study will commence in February 2013 utilising the network of 120 UK hospitals currently participating in the UK IBDGC pharmacogenetic programme (www.ibdresearch.co.uk). The collection of clinical data is aligned with the data being collected by the Royal College of Physicians UK IBD Biologics Audit. The clinical data for PANTS will be collected separately using a dedicated application held within the N3 network (www.pantsdb.co.uk). In order to avoid duplicate data entry we will share relevant anonymised data with the UK IBD Biologics Audit (and in due course with the UK IBD registry). The PANTS study aims to build a bio-resource for use by the UK IBD scientific community. Anonymised data will be made available to interested parties following appropriate ethical approval and consideration by the scientific management committee.

Patients will not be randomly allocated to one therapy or another and no attempt will be made to match populations including control for disease activity. Therefore the study has not been designed to directly compare PNR or LOR rates between IFX and ADA.

This observational study is funded by CORE, the British Society of Gastroenterology research charity and by unrestricted educational grants from Merck Sharp & Dohme (MSD) and AbbVie. The sponsor of the study is the Royal Devon and Exeter NHS Foundation Trust.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 6 years and over
* Patients with active luminal Crohn's disease involving the colon and/or small intestine (Montreal classification L1, L2 or L3), where the primary indication for anti-TNF treatment is NOT fistulising disease.
* Evidence of active disease supported by raised CRP and/or faecal Calprotectin.
* No prior exposure to anti-TNF medication.

Exclusion Criteria:

* Patient unwilling to take part.
* Unable to obtain written informed consent.
* Normal CRP and calprotectin at pre-screening.
* Patient is, in the opinion of the investigator, not suitable to participate in the study.
* Patients with contraindications to the use of anti-TNF drugs.

Ages: 6 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: UK NHS Patients with active luminal Crohn's disease.
Sampling Method: Non-Probability Sample
Enrollment: 1750 (Actual)
Dates: Start 2013-03; Primary Completion 2017-07-30 (Actual); Study Completion 2019-07-30 (Estimated)

PRIMARY OUTCOMES:
To measure the clinical, biological, genetic markers that define response to anti-TNF in patients with active Crohns disease | 3 years
  We will measure biomarkers, clinical data and genetic data through the PANTS project at multi time points.

SECONDARY OUTCOMES:
To measure the serious adverse events to Anti-TNF in Crohn's disease. | 3 YEARS
to measure the clinical, biochemical and genetic markers of durable clinical remission after anti-TNF withdrawal | 3 YEARS
To measure the clinical, biological and genetics marker for patients recruited and switched to biosimilar Infliximab (RemsimaTM and InflectraTM) including efficacy, safety and pharmacokinetics using a prospective open labelled study design. | 2 YEARS

CONTACTS AND LOCATIONS:
Overall Officials: Tariq Dr Ahmad, Principal Investigator — Royal Devon and Exeter Hospital NHS Trust
Locations (1):
- Royal Devon and Exeter Hospital NHS Foundation Trust, Exeter, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The clinical and genetic data will be entered into the Peninsular Resreach Bank or another Biobank for sharing

REFERENCES:
- [Derived] Chanchlani N, Lin S, Bewshea C, Hamilton B, Thomas A, Smith R, Roberts C, Bishara M, Nice R, Lees CW, Sebastian S, Irving PM, Russell RK, McDonald TJ, Goodhand JR, Ahmad T, Kennedy NA; PANTS Consortium. Mechanisms and management of loss of response to anti-TNF therapy for patients with Crohn's disease: 3-year data from the prospective, multicentre PANTS cohort study. Lancet Gastroenterol Hepatol. 2024 Jun;9(6):521-538. doi: 10.1016/S2468-1253(24)00044-X. Epub 2024 Apr 16. PMID 38640937
- [Derived] Bai BYH, Reppell M, Smaoui N, Waring JF, Pivorunas V, Guay H, Lin S, Chanchlani N, Bewshea C, Goodhand JR, Kennedy NA, Ahmad T, Anderson CA; UK Inflammatory Bowel Disease Pharmacogenetics Study Group. Baseline Expression of Immune Gene Modules in Blood is Associated With Primary Response to Anti-TNF Therapy in Crohn's Disease Patients. J Crohns Colitis. 2024 Mar 1;18(3):431-445. doi: 10.1093/ecco-jcc/jjad166. PMID 37776235
- [Derived] Sazonovs A, Kennedy NA, Moutsianas L, Heap GA, Rice DL, Reppell M, Bewshea CM, Chanchlani N, Walker GJ, Perry MH, McDonald TJ, Lees CW, Cummings JRF, Parkes M, Mansfield JC, Irving PM, Barrett JC, McGovern D, Goodhand JR, Anderson CA, Ahmad T; PANTS Consortium. HLA-DQA1*05 Carriage Associated With Development of Anti-Drug Antibodies to Infliximab and Adalimumab in Patients With Crohn's Disease. Gastroenterology. 2020 Jan;158(1):189-199. doi: 10.1053/j.gastro.2019.09.041. Epub 2019 Oct 7. PMID 31600487
- See also: Exeter IBD research website — http://www.ibdresearch.co.uk